CLINICAL TRIAL: NCT02889627
Title: Efficacy and Safety of Fecal Microbiota Transplantation for Epilepsy
Brief Title: Fecal Microbiota Transplantation for Epilepsy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epilepsy-CN-160816
Record Dates: First submitted 2016-08-16; First posted 2016-09-05 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2023-12

CONDITIONS: Epilepsy
Keywords: Fecal Microbiota Transplantation; Gut microbiota; Brain-gut axis; Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FMT with microbiota suspension (Experimental): Participants undergo repeated FMT with ~50ml microbiota suspension.
  Interventions: Drug: Fecal microbiota suspension

INTERVENTIONS:
Drug: Fecal microbiota suspension — The prepared microbiota suspension was infused into the participates' mid-gut or lower gut.
  Other Names: Washed fecal microbiota

SUMMARY:
Increasing evidences showed the microbiota effects on neuropsychiatric disorders. This clinical trial aims to evaluate the efficacy and safety of fecal microbiota transplantation for epilepsy.

DETAILED DESCRIPTION:
Very few literatures reported the clinical use of microbiota or bacteria for brain diseases. The most effective strategy for reconstruction of gut microbiota should be fecal microbiota transplantation (FMT). This study aims to evaluate the efficacy and safety of FMT for epilepsy. Patients were diagnosed as epilepsy by electroencephalogram (EEG) and MRI and clinical data when the study began and thent received repeated FMT with fecal from healthy donors.The antiepileptic medication regimen of patients remained unchanged after FMT. The primary outcome measure was the frequency of the seizures. Secondary outcome measure were the 50% response rate.

.

ELIGIBILITY:
Inclusion Criteria:

had been diagnosed with epilepsy for at least three months; experienced at least one seizure during the three months before WMT ;

Exclusion Criteria:

had other severe diseases, including other intestinal disorders (e.g., Clostridioides difficile infection), malignant neoplasm, cardiopulmonary failure or serious liver or kidney disease, had undergone previous FMT or WMT, had taken antibiotics within three months before starting WMT

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of the seizures | 3months
  the rates of patients who achieved a ≥50% reduction in seizure frequency from baseline to one month after WMT

SECONDARY OUTCOMES:
gut microbiota analysis | baseline, 1 week-post-FMT, 1 months-post-FMT, 3 months-post-FMT
  The stool samples of participants before and after FMT were collected and analized, by 16S rRNA and were used to investigate the crucial microbiota for devising a more efficient treatment strategy for epilepsy.
Adverse events | 3months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after FMT.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD,PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Hsiao EY, McBride SW, Hsien S, Sharon G, Hyde ER, McCue T, Codelli JA, Chow J, Reisman SE, Petrosino JF, Patterson PH, Mazmanian SK. Microbiota modulate behavioral and physiological abnormalities associated with neurodevelopmental disorders. Cell. 2013 Dec 19;155(7):1451-63. doi: 10.1016/j.cell.2013.11.024. Epub 2013 Dec 5. PMID 24315484
- [Background] Borody TJ, Khoruts A. Fecal microbiota transplantation and emerging applications. Nat Rev Gastroenterol Hepatol. 2011 Dec 20;9(2):88-96. doi: 10.1038/nrgastro.2011.244. PMID 22183182
- [Background] Cui B, Li P, Xu L, Peng Z, Xiang J, He Z, Zhang T, Ji G, Nie Y, Wu K, Fan D, Zhang F. Step-up fecal microbiota transplantation (FMT) strategy. Gut Microbes. 2016 Jul 3;7(4):323-328. doi: 10.1080/19490976.2016.1151608. Epub 2016 Mar 3. PMID 26939622